CLINICAL TRIAL: NCT05794867
Title: Comparative Study Between Use of Ultrasonic Criteria of Weaning Versus the Conventional Criteria of Weaning in Post-traumatic Acute Respiratory Distress Syndrome Patients Who Were Ventilated for a Long Time
Brief Title: Ultrasonic Weaning Criteria in Prolonged Ventilation
Status: Completed | Type: Observational
Sponsor: King Abdul Aziz Specialist Hospital (Network)
Responsible Party: Sponsor
Other Study IDs: icu- 4-23
Record Dates: First submitted 2023-03-19; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Blood Gas Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients were randomly allocated in one of two groups each group contain 100 patients.: Group A considered control group. Those patients weaned from the ventilator by the conventional criteria of weaning
  Interventions: Diagnostic Test: clinical weaning criteria
- 100 patients: group B weaned from the ventilator by the ultrasound criteria of weaning. All patients weaned from both groups followed for six days for signs of failure of weaning ,signs of post-extubation respiratory failure. And number of patients who were re-ventilated and who discharged from ICU in both groups recorded and compared.

INTERVENTIONS:
Diagnostic Test: clinical weaning criteria — Xray chest and calculation of thr rapid shallow breathing rate
  Other Names: arterial blood gases and reading on the ventilator
  Groups: Patients were randomly allocated in one of two groups each group contain 100 patients.

SUMMARY:
compare and evaluate the effect of use of ultrasonic criteria of weaning versus the conventional ways of weaning in post-traumatic acute respiratory distress syndrome (ARDS) patients who were ventilated for a long time. And compare their effect on the duration of ICU stay.

DETAILED DESCRIPTION:
It is a prospective double blind study done on total 200 patients. Who were weaned from ventilator after being ventilated for > one week due to respiratory failure. This respiratory failure was selected in our study to be from severe lung contusion and post-traumatic acute respiratory distress syndrome. Patients were randomly allocated in one of two groups each group contain 100 patients. Group A considered control group. Those patients weaned from the ventilator by the conventional criteria of weaning. While group B weaned from the ventilator by the ultrasound criteria of weaning. All patients weaned from both groups followed for six days for signs of failure of weaning ,signs of post-extubation respiratory failure. And number of patients who were re-ventilated and who discharged from ICU in both groups recorded and compared.

ELIGIBILITY:
Inclusion Criteria:

* adult patients between 18-65 years old,
* with Acute respiratory distress syndrome,
* any ventilated patients for more than one week

Exclusion Criteria:

* young or pediatric patients below 18 years.
* patients older than 65 years
* patients had Chronic Respiratory Disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — both sex are allocated randomly in one of the two groups
Study Population: It is a prospective double blind study done on total 200 patients. Who were weaned from ventilator after being ventilated for > one week due to respiratory failure. This respiratory failure was selected in our study to be from severe lung contusion and post-traumatic acute respiratory distress syndrome.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-03-19 (Actual); Study Completion 2023-03-19 (Actual)

PRIMARY OUTCOMES:
The number of patients who had no failure of weaning | 6 days
  patients followed by ultrasounds criteria

SECONDARY OUTCOMES:
The number of patients who discharged early from ICU | 6 days

CONTACTS AND LOCATIONS:
Locations (1):
- King abd el Aziz specialist hospital, Ta'if, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
the data is only laboratory data and figures read from the ventilator